CLINICAL TRIAL: NCT02174874
Title: Comparison of Ondansetron Oral Solution to Orally Disintegrating Tablets for the Management of Suspected Viral Gastroenteritis in a Pediatric Emergency Department
Brief Title: Ondansetron Oral Versus Orally Disintegrating Tablets (ODT)
Status: Completed | Type: Observational
Sponsor: Dr. Graham Thompson (Other)
Responsible Party: Sponsor-Investigator, Dr. Graham Thompson, Physician, Alberta Children's Hospital
Organization: Alberta Children's Hospital (Other)
Other Study IDs: OND - 0001
Record Dates: First submitted 2011-05-26; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Acute Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Oral Ondansetron: Arm that receive oral solution .8 mgms per ml ondansetron - Apotex Brand DIN 02291967
- Oral disintegrating tablets: Arm that receives the disintegrating tablets either 4mg or 8 mgs Glaxo Brand 4 mg DIN 02239372, 8 mg DIN 02239373

SUMMARY:
In children aged 3 months to 10 years who present to the Pediatric Emergency Department (PED) with recent, significant vomiting and moderate dehydration, is treatment with Ondansetron Orally Disintegrating Tablet (ODT) better tolerated than treatment with Ondansetron Oral Solution (OS)? Our hypothesis is that children who receive Ondansetron ODT will have 10% less vomiting within 15 minutes of administration than those receiving Ondansetron OS.

DETAILED DESCRIPTION:
Vomiting related to viral gastroenteritis is the most common presentation to the Alberta Children's Hospital Pediatric Emergency Department. Recently, a clinical pathway was implemented to improve the care and flow of patients with vomiting and/or diarrhea through the department. Administration of an antiemetic, Ondansetron, is an integral part of improving the hydration status of children managed by the pathway. However it is not know whether Oral Solution or Oral Disintegrating Tablets are better tolerated in children who have active vomiting. The investigators aim to show that children receiving Oral Disintegrating Tablets have less vomiting immediately after medication administration than children receiving Oral Solution. By demonstrating this improved tolerability the investigators will provide health care providers the stimulus for implementing Ondansetron Oral Disintegrating Tablets into their practice for children with active vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 months to 10 years with recent,
* significant vomiting and moderate dehydration who are managed according to the Alberta Health Services (Calgary and Area) Acute Childhood Vomiting & Diarrhea Pathway.
* The following definitions are used to determine inclusion according to the pathway: Recent, significant vomiting - Vomiting at least 6 episodes in the past 6 hours and at least once in the past hour; Moderate dehydration (Gorelick Score 2) - Two of the following: capillary refill time greater than 2 seconds, absence of tears, dry mucous membranes, ill general appearance.

Exclusion Criteria:

* Children who are excluded from the Alberta Health Services (Calgary and Area) Acute Childhood Vomiting & Diarrhea Pathway.
* These criteria include: Vomiting or Diarrhea for greater than 7 days, Localized abdominal pain, Chronic medical conditions affecting major organ systems (Ex, diabetes, PKU, immunodeficiency), Likely GI Obstruction (abdominal distension, bilious vomiting, absent bowel sounds), Weight less than 8kg. Children who have received anti-emetics at home will not be excluded but will be tracked.

Ages: 3 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Alberta Children's Hospital Emergency department, all patients presenting with acute gastroenteritis
Sampling Method: Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
proportion of patients who vomit within 15 minutes of administration of anti-emetic | 15 minutes
  To determine the proportion of patients aged 3 months to 10 years who present to the PED with recent significant vomiting and moderate dehydration who vomit within 15 minutes of receiving either Ondansetron Oral Solution versus Orally Disintegrating Tablets.

SECONDARY OUTCOMES:
# episodes of vomiting after ondansetron administration | While in the ED, anticipated to be on average < 5 hours
  To determine the number of episodes of vomiting while in the emergency department (after Ondansetron administration) that are experienced by the above population.
Discharged home without IV | Duration of ED visit, anticipated to be on average < 5 hours
  To determine the proportions of children in each study group that are discharged home from the Emergency Department without receiving IV fluids.

CONTACTS AND LOCATIONS:
Overall Officials: Graham Thompson, Physician, Principal Investigator — Alberta Children's Hospital, Department of Pediatrics/Medicine, University of Calgary; David W Johnson, Physician, Principal Investigator — Alberta Children's Hospital, Department of Pediatrics/Medicine, University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada